CLINICAL TRIAL: NCT03403023
Title: Corneal Tear Film Imaging of the Cornea Before and After Restasis Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, segev fani, Primary Investigator, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0178-16-MMC
Record Dates: First submitted 2018-01-11; First posted 2018-01-18 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2017-10

CONDITIONS: Dry Eye Syndrome; Tear Film Insufficiency
Keywords: Dry Eye Disease; Tear Film Imager; tear film; Cyclosporine; dry eye syndrome; keratoconjunctivitis sicca
MeSH Terms: conditions — Dry Eye Syndromes; Xerophthalmia; Keratoconjunctivitis Sicca | interventions — Cyclosporins

STUDY DESIGN:
Intervention Model Description: A single group of patients with DES is imaged before and after treatment with Restasis, a medication which is already FDA approved for this indication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DES treated patients (Experimental): This single group of patients is imaged by the Tear Film Imager (TFI) device before and after treatment with Restasis, the treatment indicated for their condition.
  Interventions: Device: Tear Film Imager; Drug: Restasis

INTERVENTIONS:
Device: Tear Film Imager — The TFI is an imaging device based on standard camera that uses white light to image the tear film in an ultra high resolution. DES patients in this study will be imaged before and 3 months after initiation of treatment with Restasis (the treatment indicated for their condition).
  Other Names: TFI
Drug: Restasis — Restasis therapy is given to all of the patients as indicated for moderate-severe DES. TFI imaging is performed before and 3 months after initiation of therapy.
  Other Names: Ophthalmic Cyclosporine A 0.05%

SUMMARY:
Dry Eye Syndrome (DES) is a disease affects the production and stability of the tear film, leading to vision disturbances and a major decrease in quality of life. The most recommended treatment for moderate-severe DES today which failed conservative therapy with lubricating eye drops is topical Cyclosporine 0.05% (Restasis®).

The Tear Film Imager (TFI) is a novel imaging modality designed for visualization of the individual tear film layers up to a resolution of 0.1 micrometers, a property not enabled by any other imaging modality for this indication to date.

In this study we wish to assess the effects of topical Cyclosporine 0.05% on the tear film using the TFI. In our previous study we found this modality yields high resolution images of the tear film, yielding significant differences between healthy and diseased (DES) eyes. We believe the TFI will improve quality of assessment and follow-up of DES patients, allowing more effective diagnosis and treatment of this disease in the future.

DETAILED DESCRIPTION:
Dry Eye Syndrome (DES) is a common eye disease that damages corneal eye surface in approximately 30% of patients who turn to treatment by Ophthalmologists. These diseases derive from changes in the quantity and quality of the tear film. Lack of timely treatment can lead to corneal surface damage, pain, infection and vision disturbances. However, effective treatment of the disease can lead to a significant improvement in patients' quality of life and improvement in visual acuity.

Conventional treatment modalities focus mainly on lubricating eye drops, but these do not treat the pathophysiologic cause which is the inflammatory process evolving on the ocular surface. Topical Cyclosporine 0.05% (Restasis®) is an anti-inflammatory drug which is the most recommended treatment option for patients with moderate-severe DES who failed conservative treatment. It has been proven to be an effective and safe treatment modality for DES patients, improving tear production, tear film stabilization and slowing disease progression.

The primary modalities for diagnosis and follow-up of DES patients today are manual and require clinician skill and experience. Moreover, current diagnosis modalities are subjective, examiner-based and are not easily reproducible. This raises the need for new diagnosis and follow-up modalities with higher resolution, precision and reproducibility qualities to allow more effective diagnosis and assessment of disease severity and well as assessment of disease progression over time.

AdOM - Advanced Optical Methods produced a Tear Film Imager, a modality based on a standard camera, using white light to image the tear film up to a resolution of 0.1 micrometers. This allows imaging of the individual tear film layers, a property currently not enabled by advanced OCT imaging modalities in use today (yielding a maximum resolution of 2.5 micrometers, thus now allowing imaging of individual tear film layers). In addition, this modality functions using full field imaging rather than raster scanned imaging, thus allowing a wide, full image of the scanned area.

The purpose of the current study is to assess the usage of the TFI in the follow-up of DES patients with moderate-severe disease treated with topical Cyclosporine 0.05%. In our previous study we found that the TFI yields high resolution tear film images, presenting significant differences between healthy and DES eyes. In this study we wish to examine the effects of topical Cyclosporine 0.05% on the tear film and assess the tear film before and after treatment. We believe this can help us better understand the effects of both the disease and the treatment on the tear film, thus allowing more effective diagnosis and treatment for future DES patients.

ELIGIBILITY:
Inclusion Criteria:

Non-pregnant adults, excluding individuals with legal misjudgement, with moderate-severe Dry Eye Syndrome (DES).

Moderate-severe DES will be defined by the following criteria:

1. Schirmer test without anesthesia < 7 mm / 5 seconds AND
2. One or more of the following (a-c):

   1. OSDI score >20
   2. Positive fluorescein staining (staining degree 1 in one of the eyes, where 0=no staining, 3=very significant staining)
   3. Tear Break-Up Time (TBUT) <= 8 seconds in one of the eyes.

Exclusion Criteria:

1. Disagreement to participate in the trial
2. Stevens-Johnson syndrome
3. Post-burn ocular injury
4. Chronic ocular diseases other that DES requiring topical treatment
5. Ocular herpes simplex disease
6. Persistent ocular inflammation or infection
7. Active blepharitis or blepharitis defined more severe than mild
8. Intraocular procedure less than 3 months prior to participation in the trial
9. Punctal plugs in one of the eyes
10. Subepithelial corneal scars
11. Neurotrophic cornea
12. Contact lens use in the 3 months prior to participation in the trial
13. Current topical treatment with Cyclosporine A
14. Previous refractive surgery
15. Keratoconus patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-01-30 (Estimated); Primary Completion 2018-05-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Tear Film changes | 3 months
  The tear film layers are imaged by the TFI before and after Restasis therapy. We will compare the differences in the tear film image in eyes before after therapy and see if there are significant differences between them.

CONTACTS AND LOCATIONS:
Overall Officials: Fani Segev, M.D., Principal Investigator — Ophthalmology department, MeirMC, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stonecipher K, Perry HD, Gross RH, Kerney DL. The impact of topical cyclosporine A emulsion 0.05% on the outcomes of patients with keratoconjunctivitis sicca. Curr Med Res Opin. 2005 Jul;21(7):1057-63. doi: 10.1185/030079905X50615. PMID 16004673
- [Background] Pflugfelder SC. Anti-inflammatory therapy of dry eye. Ocul Surf. 2003 Jan;1(1):31-6. doi: 10.1016/s1542-0124(12)70005-8. PMID 17075627